CLINICAL TRIAL: NCT04674982
Title: The Effect of Vibration on Pain During Heel Lance Procedures in Newborns
Brief Title: Vibration and During Heel Lance Procedures in Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Elif BİLSİN KOCAMAZ, Assistant Professor, University of Gaziantep
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Heel Lance Procedures
Keywords: newborns; vibration; pain; heel lance
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration Group (Experimental): In the vibration group, a vibrating device (Mini vibrator, 8.5 cm, 92-100 Hz) was applied to the middle/side area through which the sural nerve passes immediately below the knee of the extremity from which heel blood was to be collected approximately 30 seconds prior to commencement of the heel lance procedure. The vibration was continued throughout the heel lance procedure unless there was redness, swelling, bruising or a change in the skin integrity in the area to which the vibration was applied, and the vibration was stopped once the procedure was over.
  Interventions: Device: a vibrating device
- Control Group (No Intervention): No interventions were made on the newborns in the control group during the heel lance procedure.

INTERVENTIONS:
Device: a vibrating device — vibrating device (Mini vibrator, 8.5 cm, 92-100 Hz)
  Arms: Vibration Group

SUMMARY:
This study aimed to evaluate the effect of applying vibration on pain during heel lance procedures in newborns.

.

DETAILED DESCRIPTION:
Methods: This randomized, controlled, experimental study. The study sample consisted of 56 newborns determined using power analysis (vibration: 28, control:28). Newborns who underwent a heel lance procedure at the specified center, whose parents agreed to participate in the study and who had reached gestational age 38 and older were enrolled in the study. In the vibration group, a vibrating device was used for approximately 30 seconds before the heel lance procedure and continued throughout the procedure. No interventions were made on the newborns in the control group. Two nurses were employed for the heel lance procedure both for the experimental and control groups. One nurse performed the heel lance procedure for all newborns and the other nurse recorded the procedure. Pain in newborns was evaluated by the nurse who performed the heel lance procedure before the procedure, and 15-20 seconds and five minutes after the procedure, as well as by two specialists through observation of the video footage of the procedures using the NIPS. The heel lance procedure was performed by the same nurse both in the vibration and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 38 and older

Exclusion Criteria:

* Disrupted skin integrity in the device placement site, nerve damage or -deformity of the limb from which the blood would be collected,
* Genetic and congenital anomalies
* Congenital metabolic disorders,
* those who had undergone cardiopulmonary resuscitation,
* Stayed in the neonatal intensive care unit for any reason,
* Heel blood could not be collected at the first attempt,
* Osteogenesis imperfecta
* Had been given an analgesic within the preceding 6 hours

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2018-09-09 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
G Power software was used to calculate the sample size of the study. | 5 days
  G Power

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziantep University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Avan Antepli N, Bilsin Kocamaz E, Gungormus Z. The Effect of Vibration on Pain During Heel Lance Procedures in Newborns: A Randomized Controlled Trial. Adv Neonatal Care. 2022 Apr 1;22(2):E43-E47. doi: 10.1097/ANC.0000000000000918. PMID 34334677